CLINICAL TRIAL: NCT02328495
Title: Misoprostol Versus Uterine Striating by Bladder Filling for Pain Relief During Office Hysteroscopy. A Randomized Controlled Trial
Brief Title: Misoprostol Versus Uterine Striating by Bladder Filling for Pain Relief During Office Hysteroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, M.D, PhD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Misoprostol /bladder/hystero
Record Dates: First submitted 2014-12-23; First posted 2014-12-31 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Pain
Keywords: Misoprostol, Office hysteroscopy ,Pain
MeSH Terms: conditions — Pain | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Active Comparator): Misoprostol (400µg) is administered vaginally 12 hours before office hysteroscopy
  Interventions: Drug: Misoprostol
- bladder Filling (Active Comparator): Uterine straightening by bladder filling before office hysteroscopy
  Interventions: Other: Bladder Filling

INTERVENTIONS:
Drug: Misoprostol — Misoprostol (400µg) will be administered vaginally 12 hours before office hysteroscopy. A rigid 2.9 mm hysteroscope with 30° forward oblique lens and outer sheath diameter of 5 mm will be used in the procedure. The uterine cavity will be distended by warm saline at a pressure between 60-80 mmHg. All the procedures will be performed during the proliferative phase using the vaginoscopic approach as described by Betocchi and Selvaggi in 1997 . All the procedures will be diagnostic.
  Pain intensity will be assessed by visual analogue scale during the examination and 30 minutes after the procedure. A visual analogue scale ranging from 0 to 10 will be used (zero indicates no pain and 10 indicates the worst possible experienced pain).
  Arms: Misoprostol
Other: Bladder Filling — Patients in bladder filling group will be instructed to drink one liter of water and to avoid urination during the one and half hour period before office hysteroscopy procedure..A rigid 2.9 mm hysteroscope with 30° forward oblique lens and outer sheath diameter of 5 mm will be used in the procedure. The uterine cavity will be distended by warm saline at a pressure between 60-80 mmHg. All the procedures will be performed during the proliferative phase using the vaginoscopic approach . All the procedures will be diagnostic.
  Pain intensity will be assessed by visual analogue scale during the examination and 30 minutes after the procedure. A visual analogue scale ranging from 0 to 10 will be used.
  Arms: bladder Filling

SUMMARY:
The aim of this study is to compare the effectiveness of misoprostol versus uterine straightening by bladder filling for pain relief in menopausal patients undergoing office hysteroscopy.

DETAILED DESCRIPTION:
Several studies revealed that cervical ripening with misoprostol is effective in reducing pain especially in postmenopausal patients. A recent randomized controlled trial revealed that uterine striating by bladder filling prior to office hysteroscopy is associated with reduced pain perception and easier introduction of hysteroscope through the cervix.

The aim of this study is to compare the effectiveness of misoprostol versus uterine straightening by bladder filling for pain relief in menopausal patients undergoing office hysteroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal patients who have an indication for office hysteroscopy

Exclusion Criteria:

* Nulliparous patients, patients with cervical pathology and previous cesarean section or cervical surgery.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Intensity of pain [ visual analogue scale ranging from 0 to 10 ] | Pain intensity will be assessed by visual analogue scale during the procedure [an expected average of 10 minutes] and 30 minutes after the procedure

SECONDARY OUTCOMES:
Operative time | From the introduction of hysteroscope into the vagina till compilation of hysteroscopic examination[ an expected average 10 minutes]

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D,PhD, Study Chair — Cairo University
Locations (1):
- Obstetrics and Gynecology Department,Cairo university, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Celik C, Tasdemir N, Abali R, Bastu E, Akbaba E, Yucel SH, Gul A. The effect of uterine straightening by bladder distention before outpatient hysteroscopy: a randomised clinical trial. Eur J Obstet Gynecol Reprod Biol. 2014 Sep;180:89-92. doi: 10.1016/j.ejogrb.2014.06.029. Epub 2014 Jul 7. PMID 25058804
- [Derived] Fouda UM, Elshaer HS, Elsetohy KA, Youssef MA. Misoprostol versus uterine straightening by bladder distension for pain relief in postmenopausal patients undergoing diagnostic office hysteroscopy: a randomised controlled non-inferiority trial. Eur J Obstet Gynecol Reprod Biol. 2016 Aug;203:326-30. doi: 10.1016/j.ejogrb.2016.06.024. Epub 2016 Jul 1. PMID 27481125